CLINICAL TRIAL: NCT06523491
Title: Survey Data Analysis to Assess the Long-term Efficacy and Safety of Intra-articular HBISA Endoprosthesis of Synovial Fluid NOLTREX™ in Knee Osteoarthritis
Brief Title: Intra-articular Polyacrylamide Hydrogel in the Treatment of Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Research Centre BIOFORM (Industry)
Responsible Party: Sponsor
Other Study IDs: IA/PAAG-SI/OA/2021
Record Dates: First submitted 2024-06-13; First posted 2024-07-26 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: IA PAAG HBISA Hydrous biopolymer with silver ions "Argiform"
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group NOLTREX 2 courses: Group NOLTREX 2 courses consisted of 30 patients who had received 2 NOLTREX™ courses in the parent study (IA/PAAG-SI/OA/2019) and OLE (IA/PAAG-SI/OA/2020)
- Group NOLTREX 1 course: Group NOLTREX 1 course comprised 17 patients who received 1 NOLTREX™ course in the parent study (IA/PAAG-SI/OA/2019)
- Placebo group: Placebo group consisted of 10 patients who had received placebo in the parent study IA/PAAG-SI/OA/2019 and had not taken part in OLE. Of 72 patients approached, only 10 agreed to participate and completed the survey.

SUMMARY:
1-year follow-up of a randomized controlled trial with open-label extension to assess the long-term efficacy and safety of Intra-articular HBISA Endoprosthesis of Synovial Fluid NOLTREX™ in Knee Osteoarthritis.

DETAILED DESCRIPTION:
HBISA (polyacrylamide hydrogel) endoprosthesis of synovial fluid NOLTREX™ is intended for the symptomatic treatment of adult patients with osteoarthritis (OA) reducing pain and improving mobility.

The aim of this 1-year follow-up was to evaluate the long-term safety and efficacy of IA Polyacrylamide hydrogel with silver ions in patients with Kellgren-Lawrence grade 3 and 4 knee osteoarthritis who had received one or two treatment courses in the IA/PAAG-SI/OA/2019 and IA/PAAG-SI/OA/2020 studies.

Follow-up data were collected in telephone interviewing (using questionnaire) in April-July 2022, 12 months after the completion of OLE (IA/PAAG-SI/OA/2020).

ELIGIBILITY:
Inclusion criteria:

The study included patients with KL grade 2-3 knee osteoarthritis who had completed study IA/PAAG-SI/OA/2019 and IA/PAAG-SI/OA/2020.

Exclusion criteria:

Declining participation in the survey Lost to follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 57 patients divided into 3 subgroups based on treatment received:
  * Group NOLTREX™ 2 courses - 30 patients (52.63%)
  * Group NOLTREX™ 1 course - 17 patients (29.82%)
  * Placebo group - 10 patients (17.54%)
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey M Noskov, Prof. PhD, Principal Investigator — State budgetary healthcare facility of Yaroslavl Region "Clinical hospital №3"
Locations (2):
- Russia (2):
  - Private Healthcare Facilty "Clinical hospital "RZHD-Medicina" of the city Saint-Petersburg, Saint Petersburg
  - State budgetary healthcare facility of Yaroslavl Region "Clinical hospital №3", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2 NOLTREX™ Courses: Group 2 NOLTREX™ courses consisted of 30 patients who had received 2 NOLTREX™ courses in the parent study (IA/PAAG-SI/OA/2019) and OLE (IA/PAAG-SI/OA/2020).
- Group 1 NOLTREX™ Course: Group 1 NOLTREX™ course comprised 17 patients who received 1 NOLTREX™ course in the parent study (IA/PAAG-SI/OA/2019).
- Placebo Group: Placebo group consisted of 10 patients who had received placebo in the parent study (IA/PAAG-SI/OA/2019) and had not taken part in OLE
Period: Overall Study
Arm/Group | Group 2 NOLTREX™ Courses | Group 1 NOLTREX™ Course | Placebo Group
Started | 30 | 17 | 10
Completed | 30 | 17 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were described by group in the whole study population which included participants of the studies IA/PAAG-SI/OA/2020 and IA/PAAG-SI/OA/2019.
Groups:
- Group NOLTREX™ 2 Courses: Group NOLTREX™ 2 courses consisted of 30 patients who had received two NOLTREX™ courses in the parent study (IA/PAAG-SI/OA/2019) and OLE (IA/PAAG-SI/OA/2020).
- Group NOLTREX™ 1 Course: Group NOLTREX™ 1 course comprised 17 patients who received one NOLTREX™ course in the parent study (IA/PAAG-SI/OA/2019).
- Placebo Group: Placebo group consisted of 10 patients who had received placebo in the parent study (IA/PAAG-SI/OA/2019; concomitant use of paracetamol (oral NSAIDs) was allowed) and had not taken part in OLE.
- Total: Total of all reporting groups
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group | Total
Number analyzed (Participants) | 30 | 17 | 10 | 57
Age, Continuous [Mean (Standard Deviation); unit: Age in years]
  Age | 63.73 (6.55) | 61.71 (7.35) | 64.30 (7.57) | 63.23 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 10
  Male | 27 | 12 | 8 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 17 | 10 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kilogram] | 80.18 (11.87) | 75.29 (5.61) | 85.65 (12.05) | 79.68 (10.85)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.06 (3.26) | 27.04 (1.91) | 30.25 (3.09) | 28.66 (3.07)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total WOMAC Score (WOMAC-T)
Description: Mean change in the total WOMAC score from visit 1 of the parent study (baseline), visits 0 [screening] and 5 [week 23] of OLE to the end of 12-month follow-up (EOF) up to 24 months post Baseline Visit 1 Study 1. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100-mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-500 for Pain, 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales gives a total WOMAC score (0-2400), where 0 represents the best and 2400 the worst possible health status.
Time Frame: From Visit 1 Study 1 (Baseline), OLE Visit 0 (6 months post Baseline Visit 1 Study 1; coincided with Visit 5 in Study 1), OLE Visit 5 (12 months post Baseline Visit 1 Study 1) to the EOF (up to 24 months post Baseline Visit 1 Study 1)
Population: Analysis population included participants of the parent study (IA/PAAG-SI/OA/2019) and OLE (IA/PAAG-SI/OA/2020). In the study IA/PAAG-SI/OA/2019 the amount of paracetamol intake in placebo group was significantly larger compared to the NOLTREX™ group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group NOLTREX™ 1 Course: Group NOLTREX™ 1 course comprised 17 patients who received a NOLTREX™ course in the parent study (IA/PAAG-SI/OA/2019).
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
Number analyzed (Participants) | 30 | 17 | 10
score on a scale
  visit 1 study 1 | 1137.13 (375.18) | 767.47 (227.42) | 1271.60 (247.29)
  OLE visit 0 | 445.33 (252.01) | 260.29 (150.02) | 616.00 (230.18)
  OLE visit 5: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 5 | 319.07 (203.24) | 78.94 (20.77) |
  EOF | 423.00 (250.02) | 50.82 (31.78) | 722.10 (246.71)
Statistical Analysis 1: Comparison: Group NOLTREX™ 2 Courses vs Group NOLTREX™ 1 Course vs Placebo Group; No sample size calculation was performed. In the survey took part 57 patients from the parent study and OLE. The study did not have a formal hypothesis. The between-group comparison of changes from baseline (OLE visit 0) in the WOMAC-T at the end of 12-month follow-up (EOF) visit was conducted using analysis of covariance (ANCOVA) and, as a post hoc test, the Tukey test; Test type: Superiority; p = 0.00, ANCOVA — The threshold for statistical significance was p <0.05; To compare the efficacy of 1 and 2 NOLTREX courses with placebo was used ANCOVA adjusted for the baseline value with fixed factor of "treatment group"; F value = 23.31
Statistical Analysis 2: Comparison: Group NOLTREX™ 2 Courses vs Group NOLTREX™ 1 Course; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.00, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = 353.18, 95% CI 2-sided [178.91 to 527.45], Standard Error of Mean 72.27
Statistical Analysis 3: Comparison: Group NOLTREX™ 2 Courses vs Placebo Group; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.00, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -292.19, 95% CI 2-sided [-480.37 to -104.01], Standard Error of Mean 78.04
Statistical Analysis 4: Comparison: Group NOLTREX™ 1 Course vs Placebo Group; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.00, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -645.37, 95% CI 2-sided [-876.07 to -414.67], Standard Error of Mean 95.68
Statistical Analysis 5: Comparison: Group NOLTREX™ 2 Courses vs Group NOLTREX™ 1 Course vs Placebo Group; The between-group comparison of changes from baseline (study 1 visit 1) in the WOMAC-T at visit 5 was conducted using analysis of covariance (ANCOVA) and, as a post hoc test, the Tukey test; Test type: Superiority; p = 0.00, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; F value = 23.31
Statistical Analysis 6: Comparison: Group NOLTREX™ 2 Courses vs Placebo Group; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.00, Tukey's HSD; LS-means difference = -292.19, 95% CI 2-sided [-480.37 to -104.01], Standard Error of Mean 78.04
Statistical Analysis 7: Comparison: Group NOLTREX™ 1 Course vs Placebo Group; Post-hoc pairwise comparisons were performed using Tukey test; Test type: Superiority; p = 0.00, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; [LS-means difference = -645.37, 95% CI 2-sided [-876.07 to -414.67], Standard Error of Mean 95.68

2. Secondary Outcome: Change in the WOMAC Pain Score (WOMAC-A)
Description: Mean change in WOMAC-A from baseline (visit 1 [week 1] of the parent study, visits 0 [screening] and 5 [week 23] of OLE) to the end of 12-month follow-up (EOF). Patients were asked to complete the questionnaire during the study visit. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a set of standardized questionnaires used by health professionals to evaluate pain, stiffness and physical functioning of the joints in patients with knee and/or hip osteoarthritis. The WOMAC Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS. The WOMAC pain scale consists of five items: (1) walking on flat ground; (2) going up or down stairs; (3) at night while in bed; (4) sitting or lying; and (5) standing upright. The scores for the Pain subscale are summed up, with a possible score range of 0-500. Higher scores represent worse pain.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group NOLTREX™ 1 Course: Group NOLTREX™ 1 Course comprised 17 patients who received 1 NOLTREX™ course in the parent study (IA/PAAG-SI/OA/2019).
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
Number analyzed (Participants) | 30 | 17 | 10
score on a scale
  visit 1 study 1 | 233.20 (77.68) | 158.18 (63.77) | 239.10 (68.76)
  OLE visit 0 | 80.93 (50.74) | 44.24 (28.77) | 103.90 (48.31)
  OLE visit 5: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 5 | 59.70 (43.68) | 3.12 (2.87) |
  EOF | 80.27 (51.92) | 3.29 (3.74) | 131.10 (64.15)

3. Secondary Outcome: Change in the WOMAC Stiffness (WOMAC-B) Score
Description: Mean change in WOMAC-B from baseline (visit 1 [week 1] of the parent study IA/PAAG-SI/OA/2019, visits 0 [screening] and 5 [week 23] of OLE IA/PAAG-SI/OA/2020) to the end of 12-month follow-up (EOF). Patients were asked to complete the questionnaire during the study visit. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-200 for Stiffness. Higher scores represent worse stiffness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
Number analyzed (Participants) | 30 | 17 | 10
score on a scale
  visit 1 study 1 | 96.17 (38.32) | 69.94 (26.93) | 101.00 (24.51)
  OLE visit 0 | 33.23 (26.38) | 26.29 (18.11) | 56.90 (32.63)
  OLE visit 5: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 5 | 22.53 (20.70) | 21.24 (6.71) |
  EOF | 31.63 (28.20) | 7.24 (5.58) | 62.20 (28.18)

4. Secondary Outcome: Change in the WOMAC Physical Function (WOMAC-C) Score
Description: Mean change in WOMAC-C from the baseline visit 1 [week 1] of the parent study, visits 0 [screening] and 5 [week 23] of OLE to the end of 12-month follow-up (EOF). Patients were asked to complete the questionnaire during the study visit. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-1700 for Physical Function. Higher scores represent worse functional limitations. The higher the score, the poorer the function.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
Number analyzed (Participants) | 30 | 17 | 10
score on a scale
  visit 1 study 1 | 807.77 (295.02) | 539.35 (170.29) | 931.50 (182.82)
  OLE visit 0 | 331.17 (186.01) | 189.76 (109.22) | 455.20 (158.93)
  OLE visit 5: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 5 | 236.83 (146.82) | 85.59 (24.11) |
  EOF | 311.10 (175.33) | 40.29 (23.94) | 528.80 (168.15)

5. Secondary Outcome: Change in the 100-mm VAS Pain Score
Description: Mean change in the VAS pain score from the baseline visit 1 [week 1] of the parent study, visits 0 [screening] and 5 [week 23] of OLE to the end of 12-month follow-up (EOF). The visual analog scale (VAS) is one of the most commonly used measures of pain intensity. The pain VAS was self-completed by the respondent. The respondent was asked to place the slider perpendicular to the VAS line at the point that represents their pain intensity. The score was determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
Number analyzed (Participants) | 30 | 17 | 10
score on a scale
  visit 1 study 1 | 61.23 (10.90) | 64.35 (10.86) | 59.50 (10.09)
  OLE visit 0: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 0 | 20.90 (9.82) | 9.47 (5.51) |
  OLE visit 5: number analyzed (Participants) | 30 | 17 | 0
  OLE visit 5 | 20.80 (12.00) | 4.88 (3.14) |
  EOF | 28.43 (12.46) | 9.88 (13.41) | 42.70 (13.53)

ADVERSE EVENTS:
Time Frame: From visit 5 of OLE (study IA/PAAG-SI/OA/2020) to the end of follow-up study (up to 12 months) for NOLTREX Groups, and from Baseline Visit 1 Study 1 to the end of follow-up study (up to 24 months) for the Placebo Group
Description: Current study did not specifically collect adverse event data. Safety assessment was based on absolute and relative contraindications for repeated intra-articular treatment and physician-reported data, including information on analgesic intake.
Arm/Group | Group NOLTREX™ 2 Courses | Group NOLTREX™ 1 Course | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 0/30 | 0/17 | 0/10

LIMITATIONS AND CAVEATS:
Findings in the placebo group should be interpreted with caution because of the limited number of participants. Besides it should be noted that concomitant use of paracetamol was allowed in the RCT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT06523491/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT06523491/SAP_003.pdf